CLINICAL TRIAL: NCT03735108
Title: Neutrophil Extracellular Traps Mediate Antiphospholipid Antibody-induced Pregnancy Loss
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, Shihua Bao, Associate Professor, Shanghai First Maternity and Infant Hospital
Other Study IDs: ShanghaiFMIH Shihua Bao
Record Dates: First submitted 2018-11-01; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Neutrophil Extracellular Traps; Antiphospholipid Antibody-induced Pregnancy Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnancy loss group: the times of pregnancy loss more than or equal to twice
- normal control group: no history of pregnancy loss

SUMMARY:
1. Establish a multi-platform detection system for neutrophil extracellular traps in blood and tissues, and evaluate the detection performance;
2. Comparing the expression levels of neutrophil extracellular traps in peripheral blood and decidua of patients with antiphospholipid antibody-induced pregnancy loss and normal control group;
3. Comparing the expression levels of neutrophil extracellular traps in peripheral blood and decidua of mice with antiphospholipid antibody-induced pregnancy loss and normal control group;
4. After treatment of antiphospholipid antibody-induced mouse abortion model with metformin,the effect of metformin on embryo loss rate and viable embryo body weight was observed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Recurrent spontaneous abortion
* Clinical diagnosis of Antiphospholipid syndrome

Exclusion Criteria:

* Other autoimmune diseases
* Hematopoietic system diseases
* Cardiovascular system diseases
* Gastrointestinal system diseases
* Urinary system diseases
* Nervous system or mental diseases
* Have taken other drugs recently

Ages: 25 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: City
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
NETs level | through study completion, an average of 8 months
  Neutrophil extracellular traps (NETs) are networks of extracellular fibers, primarily composed of DNA from neutrophils, which bind pathogens.

SECONDARY OUTCOMES:
complete blood count (CBC) | through study completion, an average of 8 months
  CBC is a blood panel requested by a doctor or other medical professional that gives information about the cells in a patient's blood, such as the cell count for each blood cell type and the concentrations of hemoglobin.

OTHER OUTCOMES:
C3 level | through study completion, an average of 8 months
  Complement component 3, often simply called C3, is a protein of the immune system. It plays a central role in the complement system and contributes to innate immunity.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, China